CLINICAL TRIAL: NCT05626777
Title: Symptoms Control and adhErenCe Assessment During Treatment With MepolizUmab New pREfilled Devices
Acronym: SECURE
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 69HCL21_0419; 2022-501029-19-00 (Other: EU Number)
Record Dates: First submitted 2022-10-05; First posted 2022-11-25 (Actual); Last update posted 2024-11-18 (Actual); Status verified 2024-11

CONDITIONS: Asthma
Keywords: Pulmonary Medicine; severe asthma; uncontrolled; mepolizumab
MeSH Terms: conditions — Asthma | interventions — mepolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pre-filled syringe, mepolizumab 100 mg/month (Experimental): Pre-filled syringe, mepolizumab, 100 mg/month, 6 first months of treatment administered by nurse, 6 last months of treatment administered by patient
  Interventions: Drug: Pre-filled syringe, mepolizumab 100 mg/month
- Auto-injector pen, mepolizumab 100 mg/month (Experimental): Auto-injector pen, mepolizumab, 100 mg/month 12 months of treatment administered by patient
  Interventions: Drug: Auto-injector pen, mepolizumab 100 mg/month

INTERVENTIONS:
Drug: Pre-filled syringe, mepolizumab 100 mg/month — Pre-filled syringe, mepolizumab, 100 mg/month, 6 first months of treatment administered by nurse, 6 last months of treatment administered by patient
  Arms: Pre-filled syringe, mepolizumab 100 mg/month
Drug: Auto-injector pen, mepolizumab 100 mg/month — Auto-injector pen, mepolizumab, 100 mg/month 12 months of treatment administered by patient
  Arms: Auto-injector pen, mepolizumab 100 mg/month

SUMMARY:
Asthma is a common pathology, with a prevalence of 6 to 8% and more than 4 million patients in France. Its management is based on different therapeutic axes. Their use is very dependent on disease control, with therapeutic escalation, from treatment on demand to a combination of them at high dosage, according to the severe asthma's phenotype.

Despite these effective therapeutic tools, there is a lack of control of the disease in the vast majority of cases, affecting at least 60% of asthmatics. Among the factors associated with lack of control, non-compliance with inhaled therapies is frequent and requires to be systematically assessed in the absence of control.

Its evaluation by definition is complex and variously appreciated, fluctuating from 40 to 80%. The means proposed for evaluating it involve doctor/patient interviews, evaluation of the therapeutic response, questionnaires, evaluation of drug consumption (evaluation of number of empty boxes, integrated electronic device, withdrawal of drugs from pharmacies, etc).

Asthma control is commonly evaluated using the validated Asthma Control Test score, in clinical practice and/or in research fields. An ACT score greater than 20 indicates well-controlled asthma. In addition, a change of at least 3 points is likely to indicate a clinically meaningful change in asthma control (Minimally Clinical Important Difference) in an individual patient over time and a change of 4 points or more further reduces the risk that the change is due to measurement error.

In the context of severe eosinophilic asthma, Mepolizumab has shown its benefit in controlling asthma, reducing the number of exacerbations and its ability to decrease the use of oral corticosteroids (MENSA, SIRIUS).

Mepolizumab is now available in 2 new "ready-to-use" forms: a pre-filled syringe and an auto-injector pen. Both systems can be administered at home either by a nurse or by the patient himself (self-administration). The choice is left to the discretion of the prescribing pulmonologist.

These new possibilities of Mepolizumab administration offer greater freedom to the patient, possibly allowing him to empower himself by carrying out his own treatment, without constraint and without being dependent on the availability of a nurse or another healthcare professional qualified to inject Mepolizumab.

These new methods of Mepolizumab self- administration also open the field to therapeutic non-compliance, a new problem in the field of biotherapies used for the treatment of severe asthma.

The investigator hypothesize a potential therapeutic non-compliance associated with the new method of administration of Mepolizumab, with self-injection by the patient, without the assistance of a nurse.

To assess this problem, the investigator propose to compare in a therapeutic trial Mepolizumab administered by pre-filled syringe by a home nurse every month versus Mepolizumab self-administered by auto-injector pen by the patient every month.

ELIGIBILITY:
Inclusion Criteria:

1. Patient aged ≥ 18 years
2. Severe asthma diagnosed by a pulmonologist and followed for at least a year
3. Blood eosinophilia ≥ 0.15 G / L in the 12 months preceding inclusion in the trial.
4. At least 2 exacerbations in the past 12 months, each time treated with oral corticosteroid therapy or an increase in dosage of oral corticosteroid therapy prescribed for a long time, for at least 72 hours.
5. High dose inhaled corticosteroid therapy (> 800 μg / d budesonide,> 500 μg / d fluticasone,> 1000 μg / d beclometasone, etc.) and at least one second controller asthma treatment with Long-Acting Beta-Agonists or Long-Acting Muscarinic Antagonists
6. Patient must have an efficient contraception method
7. Patient affiliated to a social security scheme.
8. Patient able to give free, informed and written consent.

Exclusion Criteria:

1. Pregnant woman (urinary beta-HCG positive at inclusion) or breastfeeding
2. Active smoking or ex-smoking for less than 6 months and more than 10 pack-years
3. Exacerbation in the 4 weeks preceding first Mepolizumab injection
4. Patient who has already been treated with Mepolizumab or another anti-IL-5 or -5R treatment
5. Patient currently using a biotherapy indicated in severe asthma other than anti-IL5 or 5R treatments or stopped for less than 2 months
6. Treatment underway with another biotherapy not indicated for severe asthma
7. Patient participating in other interventional research, excluding routine care research (old regulation) and category 2 research not interfering with primary endpoint analysis
8. Other chronic respiratory pathology (bronchiectasis, chronic obstructive pulmonary disease, pulmonary fibrosis, etc.)
9. Any other uncontrolled chronic pathology, the presence of which would be considered incompatible with the performance of the study by the investigator
10. Patient under guardianship, curatorship or legal protection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2023-03-09 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Compare asthma control after 6 months of treatment between: A1 Group of patients using a pre-filled syringe administered monthly by a nurse, using a pre-filled syringe B1 Group of patients receiving self-administered monthly, using an auto-injector pen | MONTHS 6
  Proportion of patients with controlled asthma using the ACT score (asthma control test), after a period of 6 months of treatment with Mepolizumab will be compared between groups of patients.
  The ACT score is a single score varying from 5 to 25 points. Asthma is considered to be controlled when the ACT score is ≥ 20. In the study, asthma will be considered controlled if the ACT score is ≥ 20 or better controlled if it increases by at least 4 points during the treatment period.

SECONDARY OUTCOMES:
Compare asthma control a. between groups A2 and B2 (see study design §4 below for groups description) b. between groups A1 and A2 c. between groups B1 and B2 | MONTHS 12
  Proportion of patients with asthma control assessed by the ACT score between:
  1. The group of patients receiving Mepolizumab self-administered monthly, using PFS and the group of patients receiving Mepolizumab self-administered monthly using an AI from 6 months to 12 months (between groups A2 and B2)
  2. Mepolizumab administered by a PFS by a nurse for the first 6 months and self-administered by a PFS for the following 6 months in the same group of patients (between groups A1 and A2)
  3. Mepolizumab self-administered by an AI during the first 6 months and self-administered by an AI the following 6 months in the same group of patients (between groups B1 and B2).
Compare Mean change in Asthma Control Test (ACT) score in each group | months 12
  Comparison of the mean change in ACT score from baseline between groups: A1 vs B1, A2 vs B2, A1 vs A2, B1 vs B2, and A vs B
Compare the proportion of patients with an ACT score change of at least 4 points in each group | months 12
  Comparison of the proportion of patients with a change in ACT score of at least 4 points from baseline between groups: A1 vs B1, A2 vs B2, A1 vs A2, B1 vs B2, and A vs B
Compare the number of exacerbation of asthma after 6 and 12 months of treatment (between A and B) | months 12
  Comparison of the proportion of patients with an exacerbation of asthma during the 12 months of treatment (between groups A and B)
Compare the number of exacerbation of asthma requiring a visit to the emergency service or hospitalization after 6 and 12 months of treatment (between A and B) | months 12
  Comparison of the proportion of patients with an exacerbation of asthma requiring an emergency service visit or hospitalization during the 12 months of treatment (between groups A and B)
Compare the change of exacerbation of asthma before and during the 12 months of treatment between A et B | months 12
  Comparison of the proportion of patients with an exacerbation of asthma during the 12 months of treatment with Mepolizumab versus the proportion of patients with an exacerbation of asthma during the 12 months prior to treatment with Mepolizumab
Compare the proportion of patients requiring unscheduled medical consultation for asthma, after 12 months of treatment between A et B | months 12
  The proportion of patients requiring unscheduled medical consultation for asthma during the 12 months of treatment (between groups A and B)
Compare oral corticosteroids consumption before and after Mepolizumab between group A and B | months 12
  Cumulative dose of oral corticosteroids before and after 12 months of treatment with Mepolizumab (exacerbation treatment excluded) between group A and B
Compare treatment compliance between groups A and B | months 12
  Treatment compliance using the MARS-5 questionnaire administered after 6 and 12 months of treatment with Mepolizumab. The MARS-5 score will be compared between both groups of patients.
Compare bronchial inflammation by measurement of Fraction of exhaled Nitric Oxide (FeNO) after 6 and 12 months of treatment (between groups A and B) | months 12
  Carrying out a FeNO at V1, V2 and V3 after 6 and 12 months of Mepolizumab treatment between groups A and B
Compare blood eosinophilia evolution after 6 and 12 months of treatment in each grouporal corticosteroids consumption before and after Mepolizumab between group A and B | Months 0, 3, 6, 9, 12
  Performing a hemogram on peripheral blood to measure eosinophilia evolution at M0, M3, M6, M9 and M12
Compare respiratory function measurement after 6 and 12 months of treatment (between A and B) | months 1, 6 12
  First measurement : Forced Exhaled Volume 1 (FEV1) Second measurement : Forced Vital Capacity (FVC) These two measurements are volumes which will be aggregated in order to obtain one final outcome measurement : FEV1/FVC in %
Compare the safety of treatment with Mepolizumab | Months 12
  Collection of adverse events related to the study treatment throughout the study
Compare the patients' quality of life in each group | months 1, 6 12
  Calculation of the mini-AQLQ quality of life score at V1, V2 and V3
Compare the patients' quality of life in each group | months 1, 6 12
  Calculation of the SNOT-22 score at V1, V2 and V3
Compare the patient satisfaction regarding asthma treatment in each group | months 1, 6 12
  Patient satisfaction questionnaire SATQ-F at Visit 1, Visit 2 and Visit 3 and assessment of the preferences of patients in each group with respect to the Mepolizumab administration system at Visit 1, Visit 2 and Visit 3
dyspnea | months 1, 6 12
  Calculation of mMRC score at Visit 1, Visit 2 and Visit 3

CONTACTS AND LOCATIONS:
Overall Officials: Gilles Devouassoux, Pr, Principal Investigator — Departement of Pulmonology, Croix-Rousse Hospital, Hospices Civils de Lyon
Locations (8):
- France (8):
  - Service de Pneumologie CHU Besançon, Besançon
  - Service de Pneumologie CHU Dijon, Dijon
  - Service de Pneumologie et ImmunoAllergologie CHU Lille, Lille
  - Departement of Pulmonology, Croix-Rousse Hospital, Hospices Civils de Lyon, Lyon
  - Service des Maladies Respiratoires CHU Montpellier, Montpellier
  - Service de Pneumologie A APHP Bichat, Paris
  - Service des Maladies Respiratoires CHU Reims, Reims
  - Service de Pneumologie CHU Toulouse, Toulouse